CLINICAL TRIAL: NCT05987475
Title: Prospective Observational Clinical Follow-up of Euromi Biosciences Pre-filled Silicone Gel Breast Implants
Acronym: ELEGANT
Status: Recruiting | Type: Observational
Sponsor: Euromi Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: ID RCB: 2023-A00101-44
Record Dates: First submitted 2023-07-25; First posted 2023-08-14 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Breast Implant Rupture; Breast Implant; Complications
MeSH Terms: interventions — Mammaplasty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Breast reconstruction — Breast reconstruction and breast augmentation based on the indications as listed out in the instructions for use of the medical device under investigation
  Other Names: Breast augmentation

SUMMARY:
Prospective observational clinical follow-up of Euromi Biosciences silicone gel-filled breast implants - Post-market clinical investigation - ELEGANT

ELIGIBILITY:
Inclusion Criteria:

* Female;
* 18 years old and above, and under 60 years old;
* has approved and signed the informed consent form;
* eligible to receive at least one EUROMI Biosciences implant during breast reconstruction following a mastectomy or during aesthetic breast surgery;
* Willing to be followed up for a period of 10 years.

Exclusion Criteria:

* Informed pregnancy or breastfeeding at the time of inclusion
* Known hypersensitivity and / or allergy to silicone;
* Not understanding or not accepting the risks of further surgeries during follow-up;
* Body mass index > 40 kg/m²;
* Diabetes
* HbA1c levels > 7,5%;
* History of repeated failure with the implantation of similar implants;
* Tissue or fat insufficiency;
* Progressive breast cancer large tumours (>5 cm), late cancer stage and deep tumours;
* Grossly positive axillary involvement / or chest wall involvement;
* High risk of cancer recurrence;
* Tissue damage in the implant area due to irradiation of the thoracic wall;
* Pre-existing pathology in the implant area;
* General infection or infection in the implant area;
* Medical condition (poor physiological condition, psychological instability, severe smoking, obesity, coagulopathy, diabetes, severe cardiovascular or pulmonary disease, etc.) Which may, according to the judgement of the surgeon, entail excessive risk and/or post-surgical complications;
* History or presence of an autoimmune disease;
* Immunocompromised;
* History or current treatment using radiation with lower-pole scarring and thin, poorly vascularized skin/tissue / microwave diathermy / or steroids;
* Medical condition likely to interfere with her capacity to understand the follow-up requirements, to participate in the follow-up or to give her informed consent;
* Concomitantly part of another interventional clinical trial.
* Under supervision or legal guardianship
* Deprived of liberty by a judicial or administrative decision
* Not affiliated to health insurance system or is a beneficiary of such coverage

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Two groups of participants will be distinguished:
  * Group 1: Insertion of an implant in the event of a breast augmentation (for aesthetic reasons)
  * Group 2: Insertion of an implant in the event of a breast reconstruction (eg.. following breast cancer)
Sampling Method: Non-Probability Sample
Enrollment: 177 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2034-09 (Estimated); Study Completion 2034-09 (Estimated)

PRIMARY OUTCOMES:
Rate of capsular contracture | From implantation to end of study (10-year)
  To describe the rate of capsular contracture. Capsular contracture will be evaluated according to the Baker classification (from I to IV with grade III/IV considered as retractile capsular contractures).
Post-surgery rupture | From implantation to end of study (10-year)
  To describe the rate of post-surgery rupture. Rupture will be evaluated based on cases of hardening or deflation, based on clinical signs and if deemed necessary by the investigator, by medical imaging (mammography, ultrasound, MRI).

SECONDARY OUTCOMES:
Participant's QoL | From implantation to end of study (10-year)
  Quality of life: will be evaluated using the French version of the Breast Body Image Scale (BBIS).
Breast implant survival rate. | From implantation to end of study (10-year)
  Breast implant survival rate: the event will be defined as the removal of a breast implant for any reason other than participant's wish. Breast survival will be defined as the absence of breast implant removal. The analysis will be at the implant level and at the participant level, overall and by group.
Frequency of occurrence of other adverse events and complications | From implantation to end of study (10-year)
  Evaluate the frequency of occurrence of other adverse events and complications recorded during the study
Participant's and investigator's satisfaction regarding the aesthetic result | From implantation to end of study (10-year)
  Participant and investigator satisfaction with aesthetic results: questionnaire using generic 6-level Likert scale: extremely dissatisfied, very dissatisfied, somewhat dissatisfied, somewhat satisfied, very satisfied, extremely satisfied.
Reoperation rate | From implantation to end of study (10-year)
  Reoperation will be defined as a new operation at the breast implant site for any cause.
  The analyses will be performed at the implant level and at the participant level, overall and by group

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Nancy, France